CLINICAL TRIAL: NCT06392256
Title: The Influence of Soft Tissue Phenotype Modification Following Free Gingival Grafting on the Treatment of Peri-implant Mucositis
Brief Title: Effect of Free Gingival Grafting on Peri-implant Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sıla Çağrı İşler, Assoc Prof, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-21071282-050.99-630224
Record Dates: First submitted 2024-04-26; First posted 2024-04-30 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Peri-implant Mucositis; Soft Tissue Inflammation
Keywords: Peri-implant Mucositis; Keratinized Mucosa; Non-surgical Therapy; Free Gingival Graft

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PM-NS: Peri-implant mucositis-Non-surgical therapy (Active Comparator): Professional mechanical plaque removal and submarginal instrumentation using titanium curettes will be performed in the non-surgical treatment of peri-implant mucositis with KMW < 2 mm.
  Interventions: Procedure: Non surgical therapy
- PM-NS-FGG: Peri-implant mucositis-Non-surgical therapy-Free Gingival Grafting (Experimental): Professional mechanical plaque removal and submarginal instrumentation using titanium curettes will be performed in the non-surgical treatment of peri-implant mucositis with KMW < 2 mm. Free gingival grafting will be done one month after the non-surgical treatment.
  Interventions: Procedure: Non surgical therapy; Procedure: Free gingival Grafting

INTERVENTIONS:
Procedure: Non surgical therapy — Non-surgical submarginal instrumentation using titanium curettes with saline irrigation will be done once in the treatment session.
Procedure: Free gingival Grafting — In the PM-NS-FGG group, soft tissue augmentation using a free gingival graft will be performed.
  Arms: PM-NS-FGG: Peri-implant mucositis-Non-surgical therapy-Free Gingival Grafting

SUMMARY:
The goal of this randomized clinical study is to investigate the impact of soft tissue phenotype modification following free gingival grafting (FGG) in addition to the non-surgical mechanical therapy of peri-implant mucositis (PM) with keratinized mucosa width (KMW) < 2 mm over a 6-month follow-up period. Therefore, the following questions related to the study are raised:

• Does soft tissue modification following free gingival grafting around the implants with KMW < 2 mm, in addition to non-surgical mechanical therapy of PM, affect the change in bleeding on probing and the rate of complete disease resolution?

Patients who apply to the Department of Periodontology, Faculty of Dentistry, Gazi University, are systemically healthy, have implant-supported restorations installed at least one year prior to their enrollment, and are diagnosed with PM on these implants will be selected for the study. Patients with KMW < 2 mm at the respective implant sites will be treated with non-surgical mechanical treatment combined with soft tissue augmentation with FGG or non-surgical mechanical treatment alone.

DETAILED DESCRIPTION:
The primary goal of treating peri-implant mucositis (PM) is to disturb the dental implant biofilm and resolve inflammatory conditions. This aims to achieve treatment success or complete disease resolution, preventing its progression to peri-implantitis. Indeed, regardless of the non-surgical mechanical/physical instrumentation approaches and despite noticeable clinical improvements, none of the existing procedures would result in complete disease resolution [i.e., absence of bleeding on probing (BOP)] in peri-implant mucositis. Taking this into account, the execution of interventions targeted at managing modifiable risk factors plays a pivotal role in maintaining peri-implant health.

Despite the increasing evidence documenting that implant sites exhibiting either a lacking or a reduced keratinized mucosa (KM) of ≤2 mm demonstrate difficulties in eliminating bacterial biofilm, leading to inflammation around the soft tissue, the requirement for a minimum peri-implant KM width (KMW) to avoid peri-implant diseases has been a highly debated topic. Indeed, KM augmentation at implant sites with a reduced KMW has been reported to be associated with statistically significant lower plaque and gingival scores as well as peri-implant probing depths (PPD) when compared with non-augmented sites. However, there is no study evaluating primarily the effect of KM augmentation on maintaining peri-implant health and preventing peri-implant diseases.

Therefore, the aim of this study is to investigate the impact of soft tissue phenotype modification following free gingival grafting in addition to the non-surgical submarginal instrumentation of peri-implant mucositis over a 6-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

Peri-implant Mucositis

* Adult (>18 years old), systemically healthy patients,
* Presence of at least one implant affected by peri-implant mucositis characterized by the presence of bleeding on probing and/or suppuration (BoP/SoP) and the absence of bone loss beyond crestal bone level changes that occur as a result of initial bone remodeling,
* Presence of buccal peri-implant keratinized mucosa width (KMW) < 2 mm around the implants diagnosed with peri-implant mucositis,
* Patients who have implant-supported restorations installed at least one year prior to their enrollment.

Exclusion Criteria:

* Systemic diseases that could influence the outcomes of dental and surgical treatments such as uncontrolled diabetes (HbA1c > 7), active treatment phase for cancer, autoimmune diseases, osteoporosis, medications such as steroids, bisphosphonates, selective serotonin reuptake inhibitors (SSRIs), proton pump inhibitors (PPIs), and antihypertensives,
* Consumption of anti-coagulants, anti-aggregation agents, antibiotics, or corticosteroid medications during the past three months,
* Pregnancy or lactation,
* History of soft tissue grafting at the respective implant sites,
* Current untreated periodontal diseases,
* Smokers (≥ 10 cigarettes per day),
* Malpositioned implants.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Bleeding on probing (BoP) - BoP extent | 3 and 6 months after the treatment
  The number of BoP around the implants

SECONDARY OUTCOMES:
Percentage of complete disease resolution (%) | 3 and 6 months after the treatment
  The absence of BoP at more than one site per implant and deepest PPD≤5 mm.
Probing pocket depth (PPD) | 3 and 6 months after the treatment
  The distance between the bottom of the pocket and mucosal margin around the implants
Keratinized mucosa width (KMW) | 3 and 6 months after the treatment
  The distance between the peri-implant mucosal margin and the mucogingival junction and recorded to the nearest millimeter using a UNC periodontal probe
Keratinized mucosa thickness (KMT) | 3 and 6 months after the treatment
  KTT will be measured 1 mm below the mucosal margin inserting an endodontic reamer to the soft tissue, and measuring the distance between the tip of the reamer and the stopper through a digital caliper. Mucosal thickness was also categorized as thick (≥2 mm) and thin (<2 mm)
Peri-implant soft-tissue dehiscence [PISTD] | 3 and 6 months after the treatment
  The distance between the apical margin of the crown to the peri-implant mucosal margin, including exposure of the prosthetic abutment, with or without the exposure of the implant-treated surface

CONTACTS AND LOCATIONS:
Overall Officials: Sila Cagri Isler, Asso Prof, Study Director — Gazi University
Locations (1):
- Gazi University Faculty of Dentistry, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Verket A, Koldsland OC, Bunaes D, Lie SA, Romandini M. Non-surgical therapy of peri-implant mucositis-Mechanical/physical approaches: A systematic review. J Clin Periodontol. 2023 Jun;50 Suppl 26:135-145. doi: 10.1111/jcpe.13789. Epub 2023 Feb 28. PMID 36802083
- [Background] Rakic M, Tatic Z, Radovanovic S, Petkovic-Curcin A, Vojvodic D, Monje A. Resolution of peri-implant mucositis following standard treatment: A prospective split-mouth study. J Periodontol. 2024 Sep;95(9):842-852. doi: 10.1002/JPER.23-0507. Epub 2023 Dec 2. PMID 38041803
- [Background] Galarraga-Vinueza ME, Tavelli L. Soft tissue features of peri-implant diseases and related treatment. Clin Implant Dent Relat Res. 2023 Aug;25(4):661-681. doi: 10.1111/cid.13156. Epub 2022 Nov 29. PMID 36444772
- [Background] Schwarz F, Sager M, Golubovic V, Iglhaut G, Becker K. Horizontal mucosal thickness at implant sites as it correlates with the integrity and thickness of the buccal bone plate. Clin Oral Implants Res. 2016 Oct;27(10):1305-1309. doi: 10.1111/clr.12747. Epub 2016 Feb 10. PMID 26864237
- [Background] Berglundh T, Armitage G, Araujo MG, Avila-Ortiz G, Blanco J, Camargo PM, Chen S, Cochran D, Derks J, Figuero E, Hammerle CHF, Heitz-Mayfield LJA, Huynh-Ba G, Iacono V, Koo KT, Lambert F, McCauley L, Quirynen M, Renvert S, Salvi GE, Schwarz F, Tarnow D, Tomasi C, Wang HL, Zitzmann N. Peri-implant diseases and conditions: Consensus report of workgroup 4 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Clin Periodontol. 2018 Jun;45 Suppl 20:S286-S291. doi: 10.1111/jcpe.12957. PMID 29926491